CLINICAL TRIAL: NCT03806803
Title: A Multicenter Double Blind Randomized Study Comparing the Efficacy of Lyophilized Sterile Fecal Filtrate to Lyophilized Fecal Microbiota Transplantation (FMT) in the Management of Recurrent Clostridioides Difficile Infection (CDI)
Brief Title: Multicentre Blinded Comparison of Lyophilized Sterile Fecal Filtrate to Lyophilized Fecal Microbiota Transplant in Recurrent Clostridioides Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of British Columbia (Other); University of Calgary (Other); McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00087406
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Clostridia Difficile Colitis; Clostridium Difficile Diarrhea
MeSH Terms: conditions — Enterocolitis, Pseudomembranous

STUDY DESIGN:
Intervention Model Description: double blind randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: LFMT and LSFF appear identical. Randomization is performed by lab staff not involved in any aspect of treatment administration or care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LFMT (Active Comparator): Lyophilized fecal microbiota transplant capsules
  Interventions: Biological: Lyophilized fecal microbiota transplant
- LSFF (Experimental): Lyophilized sterile fecal filtrate capsules
  Interventions: Biological: Lyophilized sterile fecal filtrate

INTERVENTIONS:
Biological: Lyophilized fecal microbiota transplant — 15 capsules
  Arms: LFMT
Biological: Lyophilized sterile fecal filtrate — 15 capsules
  Arms: LSFF

SUMMARY:
Fecal microbiota transplantation (FMT) is a treatment that restores the balance of gut bacteria and is the most effective treatment for patients who suffer from recurrent Clostridioides difficile infection (CDI) brought on by antibiotic use. Although highly effective, we do not understand how FMT actually works.

Freeze-dried or lyophilized fecal microbiota transplant (LFMT) has been shown to be effective. Recently, filtered fecal slurry, free of any live bacteria, has also been shown to cure 5 such patients. The advantage of the filtered fecal slurry is that it may be safer to patients as it does not contain any live bacteria. We have conducted a pilot study comparing LFMT to lyophilized sterile fecal filtrate (LSFF) in 9 patients, and found that the success rate of treatment was 80% vs 75% in these 2 groups.

Therefore we need to perform a larger multicenter study to compare LFMT to LSFF to determine the success rate of curing these patients.

DETAILED DESCRIPTION:
This prospective double blind randomized study will enroll 248 patients with recurrent Clostridium difficile infection (RCDI) in a 1:1 ratio to receive either LFMT or LSFF by capsules.

Patients will receive 15 capsules at week 0 and be assessed at weeks 1, 4, 8 and 24. Blood, stool and urine samples will be collected. If the first treatment fails, patients will be given open label LFMT from the same donor. If treatment fails again, FMT will be offered in the form and route at the treating physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 episodes of recurrent CDI with each episode defined as 3 or more unformed stools in 24 hours associated with positive Clostridium difficile test, each occurring within 3 months of each other.
* CDI infection under symptomatic control with 3 or fewer unformed stools in 24 hours for at least 2 consecutive days prior to treatment
* Ability to provide informed consent
* Females and males must agree to effective contraception for the duration of the study

Exclusion Criteria:

* Severe or fulminant colitis
* Chronic diarrheal illnesses such as irritable bowel syndrome or inflammatory bowel disease unless under control or in remission 3 months prior to enrollment.
* Those taking or planning to take an investigational drug within 3 months of enrollment
* Chemotherapy or radiation therapy
* Oropharyngeal or significant esophageal dysphagia
* Ileus or small bowel obstruction
* Pregnant or planning to become pregnant within 3 months
* Breastfeeding or planning to breastfeed during the trial
* Active infection requiring antibiotics
* Life expectancy <6 months Those with history of total colectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Resolution of RCDI | 8 weeks
  Proportion of patients without RCDI

SECONDARY OUTCOMES:
Resolution of RCDI | 24 weeks
  Proportion of patients with sustained cure
Serious Adverse Events | 8 weeks
  Mortality directly attributable to CDI or treatment
Serious Adverse Events | 8 weeks
  Infection directly attributable to treatment
Minor Adverse Events | 1 week
  Nausea
Minor Adverse Events | 1 week
  Vomiting
Minor Adverse Events | 1 week
  Abdominal discomfort
Difficulty swallowing capsules | 1 week
  Reported by patients as ranging between none, moderate or severe
Fever | 1 week
  Temperature of >37.8C

CONTACTS AND LOCATIONS:
Overall Officials: Dina Kao, MD, Principal Investigator — University of Alberta
Locations (5):
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - University of British Columbia, Victoria, British Columbia
  - Mcgill University Health Centre, Montreal, Quebec
  - University Of Calgary, Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kao D, Wong K, Lee C, Steiner T, Franz R, McDougall C, Silva M, Schmidt TSB, Walter J, Loebenberg R, Monaghan TM, Giebelhaus RT, Harynuk JJ, Xu H, Yaskina M, MacDonald KV, Marshall DA, Louie T. Effects of lyophilised faecal filtrate compared with lyophilised donor stool on Clostridioides difficile recurrence: a multicentre, randomised, double-blinded, non-inferiority trial. Lancet Gastroenterol Hepatol. 2025 Nov;10(11):986-997. doi: 10.1016/S2468-1253(25)00190-6. Epub 2025 Sep 22. PMID 40997843